CLINICAL TRIAL: NCT02932384
Title: Passport to Wellness-Full Intervention Phase
Brief Title: Reducing HIV Risk With High Risk HIV Negative Black MSM-Passport to Wellness
Acronym: PtW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: University of California, Los Angeles (Other); University of Southern California (Other); Los Angeles Centers for Alcohol and Drug Addiction (L.A. CADA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TL13-LACA-576
Record Dates: First submitted 2016-08-30; First posted 2016-10-13 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: HIV; Men
Keywords: HIV; Black/African American; Men; Gay/bisexual; Los Angeles
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control-Passport Only (Active Comparator): Complete a needs assessment and develop a written "Passport to Wellness," an itemized set of health promoting behaviors and services aligned with lifestyle and goals. Participants are compensated based on the items they complete, services they attend.
  Interventions: Behavioral: Control-Passport Only
- Intervention-Passport and Peer Mentor (Experimental): In addition to the "Passport to Wellness" developed with project staff, study participants will select a peer mentor trained in motivational interviewing. The peer mentor will help guide the participant to complete passport items. Part of passport development will include compensation for meeting with peer mentors to form strategies for meeting goals and addressing barriers/challenges that arise.
  Interventions: Behavioral: Intervention-Passport and Peer Mentor; Behavioral: Control-Passport Only

INTERVENTIONS:
Behavioral: Intervention-Passport and Peer Mentor — In addition to the passport and incentives described below for the control condition, participants assigned to the intervention will select a peer mentor trained in motivational interviewing. The mentor will help guide the participant to complete passport items and address priorities. Participants will also be incentivized for regular meetings with his peer mentor.
  Other Names: Passport To Wellness
  Arms: Intervention-Passport and Peer Mentor
Behavioral: Control-Passport Only — A trained staff member will use a needs assessment and the participant's own priorities to develop a 'Passport to Wellness,' a personalized set of services whose access may encourage HIV prevention or address barriers to HIV testing.
  Example passport items include: getting an HIV test, attending an informational session about PEP/PrEP, meeting with a PrEP provider, attending 12-step meetings, yoga classes, a massage or Reiki session, or reviewing specific HIV prevention information online. Participants will be incentivized for each passport item they complete.
  Other Names: Control

SUMMARY:
The proposed research study will focus on Black men who have sex with men (BMSM) who

* are HIV- or unknown status AND
* have not received HIV testing in over a year or
* who test irregularly (on 9/21/2016, the protocol was changed to modify the last to criteria and focus on those who have not used PrEP in the prior six months).

and implement an innovative, culturally-informed, peer-based, and client-centered approach that is designed to increase their awareness of their HIV status and their timely entry into prevention (including PrEP), testing, care, and treatment services. The research design compares the effect of an incentives-only approach to one that uses incentives, along with the involvement of peer mentors to support timely entry into prevention, testing, care and treatment. This phase of the study is designed to assess peer-supported intervention group versus a passport/incentive-only control group over an 18-month period using a randomized trial approach.

DETAILED DESCRIPTION:
The proposed research study focuses on BMSM who have not received HIV testing in over a year, or who test irregularly, and implement an innovative, culturally-informed, peer-based, and client-centered approach that is designed to increase their awareness of their HIV status and their timely entry into prevention, care, and treatment services. On 9/21/2016, the protocol was changed to focus on those who have not used PrEP in the prior six months.

The research design compares the effect of an incentives-only approach to one that uses incentives, along with the involvement of peer mentors to support timely entry into prevention, testing, care and treatment. This phase of the study is designed to assess peer-supported intervention group versus a passport/incentive-only control group over an 18-month period using a randomized trial approach.

The Specific Aims of the full intervention phase are:

2 (Modified). To assess the effectiveness of a peer-supported, incentivized, and client-centered approach (PtW) compared to a non-peer supported, incentivized, and client-centered approach (Control) for linking at-risk BMSM to biomedical (PEP, STD testing), structural or behavioral services that support HIV prevention and care.

2a. Hypothesis: the peer-supported model (PtW) will lead to more frequent and earlier linkages to services than the non-peer supported model (Control).

2b. Hypothesis: the peer-supported model (PtW) will lead to greater reductions in HIV risk behaviors than the non-peer-supported model (Control).

3 (NEW). To assess the effectiveness of a peer-supported, incentivized, and client-centered approach (PtW) compared to a non-peer supported, incentivized, and client-centered approach (Control) for linking at-risk BMSM to PrEP services.

3a. Hypothesis: the peer-supported model (PtW) will lead to more frequent receipt of PrEP education and consultations than the non-peer-supported model (Control) 3b. Hypothesis: the peer-supported model (PtW) will lead to more frequent uptake of PrEP (defined as taking PrEP at six month follow-up) than the non-peer-supported model (Control).

ELIGIBILITY:
Inclusion criteria:

1. self identify as male
2. self-identify as Black or African American
3. sex with a male or male-to-female transgender in the last 6 months
4. intercourse without a condom in the last 6 months
5. Los Angeles County resident,
6. either is unaware of HIV status and has not tested for HIV in the last 12 months or has recently tested (within 30 days), but had not received testing in the prior 12 months

   * 6) Modified 9/21/2016 to has not taken PrEP in the prior 6 months

Exclusion criteria:

1. self-identify as female or transgender male or female
2. does not self-identify as Black or African American
3. no sex with a man or a male-to-female transgender in the last 6 months
4. no sexual intercourse in the last 6 months
5. resides outside of Los Angeles County
6. is HIV-positive OR has tested between 1 and 13 months prior to enrollment.

   * 6) Modified 9/21/2016 to has not taken PrEP in the prior 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Number self-reporting specific HIV/STD (sexually transmitted disease) Testing outcomes | 6 Months
  --Number of participants 1) human immunodeficiency virus (HIV) tested within one and six months of their baseline; 2) newly diagnosed with HIV, and 3) obtaining testing for other STDs within six months of their baseline.
Number with specific PrEP outcomes | 6 Months
  --Number of participants who attend a PrEP information session, meet with a PrEP provider, or obtain a new PrEP prescription.
Number self-reporting specific Social and Behavioral Outcomes | 6 Months
  --Number of participants who obtain social and behavioral services that support HIV prevention and care.
Percentage self-reporting specific HIV/STD (sexually transmitted disease) Testing outcomes | 6 Months
  --Percentage of participants 1) human immunodeficiency virus (HIV) tested within one and six months of their baseline; 2) newly diagnosed with HIV, and 3) obtaining testing for other STDs within six months of their baseline. Summary data may include the percentage who report HIV or STD testing.
Percentage with specific PrEP outcomes | 6 Months
  --Percentage of participants who attend a PrEP information session, meet with a PrEP provider, or obtain a new PrEP prescription. Summary items may include the percentage who report doing any of these three PrEP activities.
Percentage of self-reporting specific Social and Behavioral Outcomes | 6 Months
  --Percentage of participants who obtain social and behavioral services that support HIV prevention and care.

SECONDARY OUTCOMES:
Number of referrals HIV tested | 6 Months
  The investigators will compare between the two arms, the number of HIV tested referrals from study participants in each arm who were 1) BMSM, 2) BMSM newly diagnosed with HIV, and 3) people from other race/gender/sexual orientation groups

CONTACTS AND LOCATIONS:
Overall Officials: Nina T. Harawa, PhD; MPH, Principal Investigator — UCLA; Charles R. Drew University of Science; Ricky Bluthenthal, PhD, Principal Investigator — University of Southern California; Charles McWells, Principal Investigator — Los Angeles Centers for Alcohol and Drug Addiction (LA CADA)
Locations (2):
- United States (2):
  - Los Angeles Centers for Alcohol and Drug Abuse (LA CADA), Los Angeles, California
  - Charles Drew University of Medicine and Science, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No